CLINICAL TRIAL: NCT05931900
Title: A Prospective, Multicenter, Single Group Target Value Study for Evaluating the Safety and Effectiveness of JensClip Transcatheter Valve Repair System in The Treatment of Functional Mitral Regurgitation
Brief Title: The JensClip Transcatheter Valve Repair System for Treating Functional Mitral Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jenscare Scientific (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT-2022-07
Record Dates: First submitted 2023-06-19; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Functional Mitral Regurgitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- moderate-severe or greater (MR ≥ 3+) functional mitral regurgitation (FMR) patients (Experimental): Functional mitral regurgitation (FMR) is common in patients with myocardial infarction or dilated cardiomyopathy, and portends a poor prognosis despite guideline-directed medical therapy (GDMT).
  Interventions: Device: moderate-severe or greater (MR ≥ 3+) functional mitral regurgitation (FMR) patients

INTERVENTIONS:
Device: moderate-severe or greater (MR ≥ 3+) functional mitral regurgitation (FMR) patients — Functional mitral regurgitation (FMR) is common in patients with myocardial infarction or dilated cardiomyopathy, and portends a poor prognosis despite guideline-directed medical therapy (GDMT).

SUMMARY:
To evaluate the efficacy and safety of the JensClip transcatheter valve repair system for patients with moderate-severe or greater (MR ≥ 3+) functional mitral regurgitation (FMR) who have received adequate treatment but are still symptomatic.

DETAILED DESCRIPTION:
The clinical trial study is designed as a prospective, multicenter, single-group target-value clinical study with single-armed target value. Subjects are patients with moderate-severe or greater (MR ≥ 3+) FMR who have received adequate treatment but are still symptomatic. The safety and efficacy of the investigational product and its performance are evaluated using the above clinical trial primary endpoint and secondary endpoint indicators. All subjects in this study will be followed up at 30 days, 3 months, 6 months, and 12 months after device implantation, and clinical data obtained will be analyzed and summarized, and clinical reports will be used for submission for product registration. The study will continue to follow up subjects for 2-5 years after surgery to observe the occurrence of adverse events and to make an accurate and credible evaluation of the long-term safety and efficacy of this investigational product. All relevant clinical data will be collected, organized and statistically analyzed by an independent data management and statistics center and clinical monitoring organization. The core laboratory assesses the relevant imaging data during the clinical trial, and the CEC (Clinical Event Committee) is specially established to determine the endpoint events of the clinical trial. The clinical study consists of two phases: the first phase is a feasibility (FIM) clinical trial and the second phase is a confirmatory clinical trial; the sample size of the FIM clinical trial is not included in the second phase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with symptomatic FMR due to ischemic or non-ischemic cardiomyopathy with moderate-severe or greater mitral regurgitation (MR ≥ 3+) confirmed by echocardiography;
* Patients that have undergone adequate treatment, including treatment for conditions such as coronary artery disease, left ventricular dysfunction, heart failure, and mitral regurgitation (e.g., coronary revascularization, cardiac resynchronization therapy, and/or guideline-directed medication therapy (GDMT) at a stable dose), as judged by the local hospital heart team; Note: Any change in GDMT with ≥ 100% increase or ≥ 50% decrease in dose is considered "unstable".
* NYHA cardiac function classification ≥ Class II;
* Left ventricular ejection Fraction (LVEF) ≥ 20%;
* Left ventricular end systolic diameter (LVESD) ≤ 70 mm;
* At least one hospitalization for heart failure in the past 12 months and/or after adequate treatment, corrected BNP >150 pg/ml or corrected NT-proBNP > 600 pg/ml (correction method: If the patient has a body mass index (BMI) ≥ 20 kg/m2, BNP or NT-proBNP decreases by 4% for each 1 kg/m2 increase);
* Subjects with mitral valves anatomically suitable for mitral valve repair using this investigational device;
* Subjects who fully understand the trial protocol and purpose, voluntarily participate in the trial and sign the informed consent form, and are willing to undergo relevant examinations and clinical follow-ups.

Exclusion Criteria:

* A history of mitral valve surgery or combined valvular disease requiring surgical or interventional treatment;
* Active rheumatic heart disease, infective endocarditis;dian
* Patients diagnosed with hypertrophic cardiomyopathy, restrictive cardiomyopathy, infiltrative cardiomyopathy (e.g., amyloidosis, hemochromatosis), constrictive pericarditis;
* Left intracardiac masses, bulges, thrombi and/or mitral valve leaflets, tendinopathy indicated by imaging;
* Severe chronic obstructive pulmonary disease (COPD) requiring continuous home oxygen therapy or long-term steroid hormone medication;
* Severe right heart insufficiency or pulmonary hypertension (pulmonary artery systolic pressure > 70 mmHg measured by ultrasound or right heart catheter; if measured at the same time, the right heart catheter measurement shall prevail);
* Patients who have had an acute myocardial infarction, stroke/transient ischemic attack (TIA) and/or gastrointestinal bleeding within 30 days; Patients who have undergone any transcatheter cardiovascular intervention, carotid artery surgery, pacemaker implantation, cardiac resynchronization therapy (CRT-P, CRT-D) or implantable cardioverter defibrillator (ICD) within 30 days, or cardiovascular surgery within 180 days;
* Hemodynamic instability, with systolic blood pressure < 90 mmHg in the absence of afterload-reducing drugs, or cardiogenic shock or the need for vasoactive drugs, intra-aortic balloon pump, left ventricular assist devices, etc.;
* Patients with known bleeding disorders, coagulation disorders, and/or clear contraindications to the use of anticoagulants and antiplatelet agents;
* Known hypersensitivity to product composition;
* Patients with clear contraindications to transesophageal echocardiography, contraindications to tracheal intubation, and/or the presence of contraindications to general anesthesia;
* Modified Rakin score ≥ 4;
* Patients with a life expectancy of < 12 months or who have undergone a heart transplant or are scheduled to have a heart transplant within 12 months after surgery;
* Patients who are enrolled in other drug or device clinical trials and have not completed follow-up of the primary endpoint;
* Pregnant or breastfeeding women or those planning to become pregnant within the next 12 months;
* Other conditions that the investigator considers inappropriate to participate in this clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality or hospitalization rate | 12 months
  All-cause mortality or hospitalization rate for heart failure 12 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Fuwai Cardiovascular Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No